CLINICAL TRIAL: NCT05674955
Title: Circuit Weight Versus Aerobic Training on Selected Cardiovascular Indices and Functional Capacity in Patients With Ischemic Cardiomyopathy.
Brief Title: CWT Versus AT on Selected Cardiovascular Indices and Functional Capacity in Patients With Ischemic Cardiomyopathy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Samira Shukrey Shaffik Eshak, Domenstrator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Cw versus AT in cardiomyopathy
Record Dates: First submitted 2022-12-10; First posted 2023-01-09 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Ischemic Cardiomyopathy

STUDY DESIGN:
Intervention Model Description: 3 groups of ischemic cardiomyopathy patients. 1st group receive circuit weight training. 2nd group receive aerobic. 3rd group receive medications
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Circuit weight group (Experimental)
  Interventions: Diagnostic Test: Circuit weight versus aerobic training
- Aerobic group (Experimental)
  Interventions: Diagnostic Test: Circuit weight versus aerobic training
- Control Group (Experimental)
  Interventions: Diagnostic Test: Circuit weight versus aerobic training

INTERVENTIONS:
Diagnostic Test: Circuit weight versus aerobic training — Circuit weight :Duration: 30 min-60 min (total session) Frequency: 3 times / week. Intensity: increased load was established when subject was able to complete 12 repetitions ( Wayne, 2014)
  B- Aerobic training:
  This mode of exercise will be conducted for study group B as follows:
  Intensity: started by 60-85% of target heart rate according to each patient response Target heart rate (THR) = 60% -85% (maximum heart rate-resting heart rate) + resting heart rate Maximum heart rate (MHR) = (220-Age). Mode: Walking on treadmill. Duration: Each session consisted of 10 minutes warming up firstly then 30 minutes time of session ended by 10 minutes cool down exercises.
  Frequency: Three times / week (Nishi et al., 2011).
  C-Traditional medical treatment:
  This treatment will be conducted for all group A, B and C.

SUMMARY:
To compare between the effect of circuit weight and aerobic training on selected cardiovascular indices and functional capacity in patients with ischemic cardiomyopathy.

DETAILED DESCRIPTION:
Ischemic cardiomyopathy (ICM) is a term that refers to the heart's decreased ability to pump blood properly due to myocardial damage brought upon by ischemia. Ischemic cardiomyopathy has a spectrum of clinical changes which eventually leads to congestive heart failure (CHF). Initially, there is a reversible loss of cardiac contractile function because of decreased oxygen supply to the heart muscle; however, when there is ischemia for a prolonged period, there is irreversible cardiac muscle damage resulting in cardiac remodeling. Remodeling is primarily achieved by myocardial fibrosis which results in decreased cardiac function, arrhythmia, and possible cardiac conduction system impairment. In ischemic cardiomyopathy, there is a significant impairment of the left ventricular systolic function, with a left ventricular ejection fraction (LVEF) less than 40% (Bhandari et al., 2021).

ELIGIBILITY:
Inclusion Criteria:

* Sixty male patients with ischemic cardiomyopathy as a result of a recent acute myocardial infarction event (≤2 months) with 40%<LVEF<50%.
* They are functionally classified as class II according to New York Heart Association (NYHA).
* Their age will be ranged from 45 to 55 years old.
* Their BMI will be ranged from 25 to 29.9 kg/m².
* They will have good mentality.

Exclusion Criteria:

* Recurrent coronary heart disease.
* Severe valvular diseases.
* Underlying pulmonary disease (aspiration pneumonia, chronic obstructive pulmonary disease, pneumothorax, etc.).
* Inability to ambulate owing to physical problems (paresis induced by cerebral stroke, spinal cord injury, amputation, severe pain, dyspnea, etc.).
* muskloskletal problems (e.g. severe osteoarthritis or ankylosing spondylitis).
* Impaired cognitive function (vascular dementia, Alzheimer's dementia, other psychological disease, etc.)

Ages: 45 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-08-25 (Actual); Primary Completion 2024-10-25 (Actual); Study Completion 2024-10-25 (Actual)

PRIMARY OUTCOMES:
Ejection fraction | 2 months
  Will be measured by precentge

SECONDARY OUTCOMES:
Blood pressure | 2 months
  Will be measured by mmhg

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Giza, Egypt

REFERENCES:
- [Background] Nishi I, Noguchi T, Iwanaga Y, Furuichi S, Aihara N, Takaki H, Goto Y. Effects of exercise training in patients with chronic heart failure and advanced left ventricular systolic dysfunction receiving beta-blockers. Circ J. 2011;75(7):1649-55. doi: 10.1253/circj.cj-10-0899. Epub 2011 May 25. PMID 21613745